CLINICAL TRIAL: NCT04828863
Title: Neurocognitive Outcomes and Quality of Life in Adults With Maple Syrup Urine Disease (MSUD)
Status: Completed | Type: Observational
Sponsor: Children's Hospital of Philadelphia (Other)
Responsible Party: Sponsor
Other Study IDs: 21-018443
Record Dates: First submitted 2021-03-24; First posted 2021-04-02 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-06

CONDITIONS: Maple Syrup Urine Disease
MeSH Terms: conditions — Maple Syrup Urine Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Index subjects: 25 young adults with MSUD who are 21 years and older.
  Interventions: Behavioral: Neurocognitive testing
- Control subjects: 25 age-matched siblings or acquaintances who do not have MSUD and are 21 years and older
  Interventions: Behavioral: Neurocognitive testing

INTERVENTIONS:
Behavioral: Neurocognitive testing — Participants will undergo a battery of neurocognitive tests that examine intellectual, executive, and adaptive function. The tests will be given remotely via internet-based surveys.

SUMMARY:
Maple Syrup Urine Disease (MSUD) is a disorder of protein metabolism that leads to neurological differences. It is an exciting time where people diagnosed with MSUD are living longer. The investigators want to learn about how adults with MSUD think, feel, and live. The purpose of this research study is to 1) look at thinking skills, behavior skills, life skills, and quality of life in adults with MSUD and 2) measure how medical and personal factors impact these areas. The results of the study will be used to learn how to best help adults with MSUD and how to prepare for their success. In this study, the participants will answer questions on thinking, life skills, behavior skills, and quality of life. These questions will be completed on the internet. The participants will have a formal testing of their thinking and behavior completed virtually. The participants may also have a 1-2-hour telephone conversation about their life. All tests will occur virtually at home. The investigators will send the participants a letter with the results of thinking and behavior tests.

ELIGIBILITY:
Inclusion Criteria for Index Subjects:

* Males or females 21 years and older
* Diagnosis of MSUD
* Ability to communicate verbally or using augmentative communication effectively to participate in appropriate neurocognitive testing

Inclusion Criteria for Comparison Subjects:

* Males or females 21 years and older
* Sibling or acquaintance of index subject
* Ability to communicate verbally or using augmentative communication effectively to participate in appropriate neurocognitive testing

Exclusion Criteria for all subjects:

* Inability to communicate verbally or using augmentative communication effectively to participate in appropriate neurocognitive testing
* Subjects or guardians or who, in the opinion of the Investigator, may be non-compliant with study schedules or procedures.
* Subjects or guardians who do not have internet access
* Subjects who do not speak English as a primary language

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population will include 25 adults with MSUD and 25 age-matched adults for the comparison group.
Sampling Method: Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2021-06-12 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
Neurocognitive Outcome: Executive Function | 1 year
  The Behavior Rating Inventory of Executive Function for Adults will be completed, scored, and standardized to age-matched norms.
Neurocognitive Outcome: Adaptive function | 1 year
  The Adaptive Behavior Assessment System 3 (ABAS-3) will be completed, scored, and scaled to age-matched norms.
Neurocognitive Outcome: Executive Function | 1 year
  The Adaptive Cognitive Evaluation will be completed, scored, and standardized to age-matched norms.

SECONDARY OUTCOMES:
Health-related Quality of Life | 1 year
  The World Health Organization Quality of Life-BREF quality of life scale will be completed by self-report and informant repot. This report will be scored and scaled to the age-match comparison group. Scores range from 0-100 with higher scores correlating with better outcome.
Transition to adult-centered healthcare | 1 year
  Readiness for transition to adult-centered healthcare will be assessed using the • Transition Readiness Assessment Questionnaire (TRAQ) self-report and informant report. This report will be score.

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Gold, MD, PhD, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared.